CLINICAL TRIAL: NCT01789099
Title: A Phase I/IIa Study of UV1 Vaccination in Patients With Non Small Cell Lung Cancer.
Acronym: UV1-hTERT2012L
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ultimovacs ASA (Industry)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-001852-20
Record Dates: First submitted 2013-02-08; First posted 2013-02-11 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer; Peptide vaccine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UV1 synthetic peptide vaccine and GM-CSF (Experimental): GM-CSF (Leukine) followed by UV1 peptide vaccine with escalating concentrations (100, 300 and 700 microgram) will be injected intradermally in the lower abdomen.
  Interventions: Biological: UV1 synthetic peptide vaccine and GM-CSF

INTERVENTIONS:
Biological: UV1 synthetic peptide vaccine and GM-CSF
  Other Names: UV1; Leukine

SUMMARY:
In this study, up to 21 patients with lung cancer will receive UV1 (a therapeutic synthetic peptide vaccine) at different dose levels. The safety and tolerability of UV1 as well as immunological response will be assessed. The purpose of this study is to select a biological dose of peptides for further clinical trials. Study recruitment completed at 6 patients in every dose level.

The main study treatment phase of this study is completed and will be reported separately.

Follow-up is ongoing

DETAILED DESCRIPTION:
This is an open label dose-escalating phase I/IIa study of UV1 peptide vaccination in patients with NSCLC after completion of radiation therapy and/or chemotherapy. Patients will be enrolled in this study if they have achieved complete response (CR), partial response (PR) or stable disease (SD) at least 4 weeks after completion of standard first line therapy.

The following 2-step design will be used:

1. Conventional dose escalation with at least 3 patients per dose level (3 selected dose levels).
2. Expansion of each dose level to a total of 6 patients for assessment of immune response levels.

13 UV1 vaccinations will be given during the first 6 months (week 26) of treatment, unless clinical deterioration or unacceptable toxicity is encountered. Granulocyte-macrophage colony-stimulating factor (GM-CSF) (Leukine ®) will be used as adjuvant for 11 of the 13 doses of UV1.

After completion of the main study treatment period at week 26, if the patient agrees, additional vaccinations may be considered for the following patients:

* Immune responders within first 6 months
* Immune non-responders providing they have at least SD

ELIGIBILITY:
Inclusion Criteria:

* Patient with Non Small Cell Lung Cancer (NSCLC) who has been treated with palliative radiotherapy and/or at least three courses of chemotherapy, and has achieved stable disease (SD), partial response (PR) or complete response (CR) confirmed by CT scan at least 4 weeks after end of treatment. Previous curative radiotherapy is allowed as long as the patient has relapsed and received palliative chemotherapy.
* No evidence of disease progression at the time of inclusion
* Must be ambulatory with an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Must be at least 18 years of age.
* Must have lab values as follows:
* White Blood Cells ≥ 1.5 x 109/L
* Platelets ≥ 100 x 109/L
* Hemoglobin ≥ 9g/dL (≥ 5.6 mmol/L)
* Creatinine ≥ 140 µmol/L
* Bilirubin < 20% above the upper limit of normal
* ASAT and ALAT ≤ 2.5 the upper limit of normal
* Albumin ≥ 2.5 g/L
* Signed informed consent

Exclusion Criteria:

* History of other prior malignancy, with the exception of curatively treated basal cell or squamous cell carcinoma of the skin, cervical cancer stage IB or effectively treated malignancy that has been in remission for over 5 years and is highly likely to have been cured.
* Treatment with any other investigational medicinal product (IMP) within 4 weeks prior to first administration of study drug.
* Adverse reactions to vaccines such as anaphylaxis or other serious reactions.
* History of immunodeficiency or autoimmune disease such as rheumatoid arthritis, systemic lupus erythematosus, sclerodermia, polymyositis-dermatomyositis, juvenile onset insulin-dependent diabetes, or a vasculitic syndrome.
* Significant cardiac or other medical illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, or serious cardiac arrhythmia.
* Known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may however participate provided they meet the following criteria:

  1. Inactive metastases (without evidence of progression which is documented by CT or MRI within 4 weeks prior to the planned study treatment date), and
  2. If prednisolone or equivalent treatment is required; no more </=10mg/day is permitted.
* Active infection requiring antibiotic therapy.
* Pregnancy or lactation.
* Woman of childbearing potential not using any reliable and adequate contraceptive methods defined as use of oral, implanted, injectable, and mechanical or barrier products for the prevention of pregnancy.
* Known hypersensitivity to any of the components of the vaccine
* Known hypersensitivity to Leukine®, yeast derived products or any component of the product
* Patients who test positive for hepatitis B, C or HIV.
* Any other anti-tumor treatment within 4 weeks of study entry (including chemotherapy, immunotherapy, endocrine therapy, cytokines, interferons, protease inhibitors and gene therapy).
* Use of not permitted concomitant medication:
* chronic corticosteroids except for asthma inhalers / topical use
* any agent with a known effect on the immune system, unless it is being given at dose levels that are not immunosuppressive, e.g. prednisone at 10mg/day or less.
* any alternative and complementary drugs that may affect the immune system or be potentially harmful to patients participating in phase I studies.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-04-08 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability of UV1. | up to 2 years and 3 months.
  Frequency and severity of adverse events and serious adverse events. Biochemistry and hematology results, vital signs and ECOG performance status will be assessed.
Immunological response | Up to 2 years and 3 months.
  Number of T-cell responses including time to T-cell responses (up to 6 months), level of response and duration of response.

SECONDARY OUTCOMES:
Assessment of anti tumor activity | Up to 2 years and 3 months
  Tumor response and progression free survival (PFS)
Selection of biological dose of peptides for further clinical trials. | Up to 2 years and 3 months
  Safety profile and immunological responses of each dose level.

OTHER OUTCOMES:
Potential correlation between human cytomegalovirus status and immune response | Up to 2 years and 3 months
  Determination of human cytomegalovirus (CMV) status
Further characterization of the immune reaction triggered by the treatment. | Up to 2 years and 3 months
  Extended immunological analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Paal F. Brunsvig, MD PhD, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Brunsvig PF, Guren TK, Nyakas M, Steinfeldt-Reisse CH, Rasch W, Kyte JA, Juul HV, Aamdal S, Gaudernack G, Inderberg EM. Long-Term Outcomes of a Phase I Study With UV1, a Second Generation Telomerase Based Vaccine, in Patients With Advanced Non-Small Cell Lung Cancer. Front Immunol. 2020 Nov 26;11:572172. doi: 10.3389/fimmu.2020.572172. eCollection 2020. PMID 33324397